CLINICAL TRIAL: NCT05456711
Title: Investigation of the Relationship Between Femoral Cartilage Thickness and Inflammatory Parameters, Pain Severity and Functionality in Knee Osteoarthiritis
Brief Title: Femoral Cartilage Thickness in Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2022.05.103
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- knee osteoarthritis: ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality
  Interventions: Diagnostic Test: ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality
- healthy control: ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality
  Interventions: Diagnostic Test: ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality

INTERVENTIONS:
Diagnostic Test: ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality — ultrasonographic measurement for femoral cartilage thickness VAS for pain severity WOMAC for functionality

SUMMARY:
The aim of the study to investigate the relationship between femoral cartilage thickness in Ultrasonographic evaluation and inflammatory parameters, pain severity and functionality in participants with Knee Osteoarthritis

DETAILED DESCRIPTION:
Aim: The aim of the study is to investigate the relationship between femoral cartilage thickness and inflammatory parameters, pain severity and functionality in participants with Knee Osteoarthritis.

Methods: This study is designed as a prospective, cross-sectional trial. 90 participants aged between 50-65 years with knee osteoarthritis(OA) and at least 50 participants without any symptom for knee OA are included in the study in accordance with the inclusion criteria. Participants' demographic characteristics will be evaluated, and ultrasonographic measurement will be performed for measuring femoral cartilage thickness. Visual Analog scale will be used for pain severity and Western Ontario and McMaster Universities Osteoartrit index (WOMAC) will be used for assessing functionality of the patients. Also hematologic parameters(neutrophils, leucocytes, lymphocytes, platelet, CRP, erythrocyte sedimentation rate) will be evaluated for investigating the inflammation. The relationship between femoral cartilage thickness and inflammatory parameters, pain severity and functionality in knee osteoarthritis will be analysed for both group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as knee osteoarthritis
* aged between 50-65 years
* volunteer to participate in the study

Exclusion Criteria:

* limitation of cooperation
* moderate to severe dementia or mental retardation, which may cause limitations in examination, testing and treatment
* refusal to participate in the study
* pprevious total knee prosthesis surgery
* secondary osteoarthritis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged between 50-65 years, female and male, diagnosed as knee osteoarthritis for study group and having no symptoms for knee OA for control group
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
ultrasonography | 1 day
  measurement of femoral cartilage thickness
Visual Analog Scale | 1 day
  evaluation of pain severity
Western Ontario and McMaster Universities Osteoarthritis Index | 1 day
  evaluation of functionality
neutrophil account | 1 day
  neutrophil account
lymphocyte account | 1 day
  lymphocyte account
monocyte account | 1 day
  monocyte account
platelet account | 1 day
  platelet account
eritrocyte sedimentation rate | 1 day
  eritrocyte sedimentation rate
C-reactive protein | 1 day
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Merve D. Korkmaz, M.D., Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided